CLINICAL TRIAL: NCT00673907
Title: Health Effects Related to Exposure to Particle Pollution From Woodburning
Brief Title: HIPWOODS - Health Effects Related to Exposure to Particle Pollution From Woodburning Stoves
Acronym: HIPWOODS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: University of Copenhagen (Other); Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 2104-05-0003; Projekt nr: 0502-
Record Dates: First submitted 2008-05-05; First posted 2008-05-07 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-02

CONDITIONS: Airway Inflammation; Systemic Inflammation
Keywords: Wood smoke; Health effects; Human; Airway inflammation; Cardiovascular effects

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Sham Comparator): Clean air
  Interventions: Other: Wood smoke particles
- 2 (Experimental): Wood smoke particle concentration of 200 ug/m3
  Interventions: Other: Wood smoke particles
- 3 (Experimental): Wood smoke particle concentration of 400 ug/m3
  Interventions: Other: Wood smoke particles

INTERVENTIONS:
Other: Wood smoke particles — Subjects are exposed at rest to the exposures for 3 h in our climate chamber

SUMMARY:
The study intends to focus on health effects and symptoms related to particle exposure from wood burning stoves

The objective is to determine whether moderate exposure to particles from wood smoke in a real life situation causes an systemic inflammatory response in peripheral blood or in lower airways. 24 healthy subjects (normal healthy subjects and mild asthmatics to study the asthmatic response) is selected for the study. A randomized double blind crossover procedure will be followed with a PM exposure concentration of 200ug/m3, 400ug/m3 or clean air as the control exposure. Exposure will take place in a climate chamber using wood burning in an appropriate wood stove.

DETAILED DESCRIPTION:
Public health is concerned with the physical, mental and environmental health of communities and populations at risk for disease and injury. Generally, the determination of health effects associated with indoor and outdoor exposures is difficult since documented cause-and-effect relationships are rare and the exposure and dosage data is sparse. Information about actual human exposure to different types of pollution has several important uses, including informing risk assessments, helping predict the potential consequences of exposures, and developing exposure criteria for regulations and other public policy guidance.

Wood-burning stoves have been a popular heating source for decades. Unfortunately, wood-burning stoves can emit substantial quantities of pollutants to outdoor and indoor air. Among the pollutants are: chlorinated dioxin, carbon monoxide, methane, volatile organic compounds (VOC), nitrogen oxides, polycyclic aromatic hydrocarbons (PAH), and fine particulate matter (PM10, PM2.5, fine and ultra fine particles). Recent studies indicate that the use of wood-burning stoves for heating of dwellings is one of the important outdoor particle sources [Glasius et al. 2004] in residential district in Denmark. This has resulted in an increase in public exposure to indoor and outdoor wood smoke related pollutants, which has prompted widespread concern about the adverse human health consequences that may be associated with wood smoke exposure.

Air pollution is a major aggravation of respiratory symptoms and disease. Effects are decreases in pulmonary function and evidence of inflammation as well as suggestions of increases in chronic respiratory disease. Orozco-Levi et al. (2006) showed strong association between wood smoke exposure and obstructive pulmonary disease. Several studies have shown that especially the small particles, has an effect on airways, and that asthmatic subjects may be the group at greatest risk from air pollutants. The awareness of the impact of airborne particles, particularly fine and ultra fine particles, on health is growing. In recent years, exposure to fine and ultra fine airborne particles has been identified as an important factor affecting human health [Seaton et al., 1995; Schwartz et al., 1996; Oberdörster et al., 1994; Alvin et al., 2000]. Several researchers hypothesize that an increased mortality is associated with the particle levels prevailing in urban air [Jamriska et al., 1999; Dockery et al., 1993]. Mølhave et al (2000; 2005) have suggested that reactive short-lived compounds resulting from reactions between ozone and particulate matter cause indoor air quality complaints and objective health effects such as impaired lung functions.

Particulate air pollution is also known to increase cardiovascular morbidity and mortality. Still the existing scientific knowledge and foundation for evaluating the underlying mechanisms and influence of particle exposure on human immune system are limited. Wood smoke particles, at levels that can be found in smoky indoor environments, seem to affect inflammation. Barregard et al observed a significant increase in S-Amyloid and Faktor VIII/vWf after 0, 3 and 20 hours of exposure to wood smoke. After 20 hours also and increase in Faktor VIII was registred. Surpise-lingly, an IL.-6 decrease was observed after 3 hours. [Barregard et al, 2006]. The particles may also act by increasing blood coagulation factors [Seaton et al 1995]. Both effects may be involved in the mechanisms whereby particulate air pollution affects cardiovascular morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Twenty-four, non-smoking atopic volunteers with normal lung function and bronchial reactivity are recruited for the study. Atopy is determined by skin-prick testing to common aeroallergens.

Exclusion Criteria:

* Smokers, pregnant women and other subjects with current or previous diseases, which could involve a risk for the subject or possibly influence the outcome measurements, will be excluded from the study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2007-01; Primary Completion 2008-06 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Different Inflammation Biomarkers | Baseline and follow up measurement after exposure 0 hours post, a 6 hours post and 20 hours post.

SECONDARY OUTCOMES:
Baseline and follow up measurements are: spirometry, exhaled breath condensate, nasal lavage, nasal patency, blood sampling and symptoms. | Baseline and follow up measurement after exposure 0 hours post, a 6 hours post and 20 hours post.

CONTACTS AND LOCATIONS:
Overall Officials: Torben Sigsgaard, Professor, Principal Investigator — Department of Environmental and Occupational Medicine , Institute of Public Health , The Faculty of Health Sciences
Locations (1):
- Institute of Environmental and Occupational Medicine , Institute of Public Health , The Faculty of Health Sciences, Aarhus C, Denmark